CLINICAL TRIAL: NCT01760408
Title: SustainTM,LLC: A.S.P.E.N.'s National Patient Registry for Nutrition Care- Home Parenteral Nutrition
Brief Title: Sustain, A.S.P.E.N. HPN Registry 2011
Status: Completed | Type: Observational
Sponsor: Sustain, LLC of the American Society for Parenteral and Enteral Nutrition (Other)
Responsible Party: Sponsor
Other Study IDs: SustainHPN2011
Record Dates: First submitted 2012-12-31; First posted 2013-01-04 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Patients Requiring Home Parenteral Nutrition

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Home PN - pediatric: Pediatric patients (under 18) on Home PN
  Interventions: Other: all patients on Home Parenteral Nutrition
- Adult patients on Home PN: Adult patients on Home PN
  Interventions: Other: all patients on Home Parenteral Nutrition

INTERVENTIONS:
Other: all patients on Home Parenteral Nutrition

SUMMARY:
The American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.) developed a Web-based registry for nutrition care launched in early 2011, initially focusing on the home parenteral nutrition (HPN) patient population. The purpose of Sustain is to collect information regarding the patients and populations who require HPN in the United States, measure outcomes associated with HPN, allow institutional benchmarking against the aggregate data, and publish the findings to improve the quality of care for patients receiving HPN. The registry is open to all sites (hospital and home based) who care for new or existing HPN patients.

ELIGIBILITY:
Inclusion Criteria:must receive PN at home -

Exclusion Criteria:patients receiving PN in long-term care or as IDPN

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients receiving parenteral nutrition at home
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
catheter infection rate | per 1000 PN days
  catheter infection rate normalized per 1000 PN days

SECONDARY OUTCOMES:
rehospitalization rate | ongoing
  rehospitalization rate per 1000 PN days

CONTACTS AND LOCATIONS:
Locations (1):
- A.S.P.E.N., Silver Spring, Maryland, United States

REFERENCES:
- [Background] Guenter P, Robinson L, DiMaria-Ghalili RA, Lyman B, Steiger E, Winkler MF. Development of Sustain: A.S.P.E.N.'s National Patient Registry for Nutrition Care. JPEN J Parenter Enteral Nutr. 2012 Jul;36(4):399-406. doi: 10.1177/0148607111432760. Epub 2012 Jan 26. PMID 22282869
- [Result] Winkler MF, DiMaria-Ghalili RA, Guenter P, Resnick HE, Robinson L, Lyman B, Ireton-Jones C, Banchik LH, Steiger E. Characteristics of a Cohort of Home Parenteral Nutrition Patients at the Time of Enrollment in the Sustain Registry. JPEN J Parenter Enteral Nutr. 2016 Nov;40(8):1140-1149. doi: 10.1177/0148607115586575. Epub 2015 May 13. PMID 25972431